CLINICAL TRIAL: NCT00113048
Title: A Phase I Study of Subcutaneously Administered CAMPATH in CD52 Expressing Hematologic Malignancies
Brief Title: Subcutaneously Administered CAMPATH in CD52 Expressing Hematologic Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM111
Record Dates: First submitted 2005-06-03; First posted 2005-06-06 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Hematologic Malignancies
Keywords: CD52 Expressing Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Alemtuzumab

INTERVENTIONS:
Drug: CAMPATH (alemtuzumab)

SUMMARY:
This phase I study will involve escalating doses of CAMPATH until the goal dose for the cohort is tolerated. The CAMPATH goal dose will be administered to the patient subcutaneously (SQ) 3 times per week for up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or refractory hematologic malignancy. The anticipated patient population are patients with chronic lymphocytic leukemia (CLL), non-Hodgkin's lymphoma or myeloma
* Patients with a history of a hematologic malignancy that has previously been shown by flow cytometry or immunophenotyping analysis to express CD52
* Any chemotherapy, major surgery or irradiation must have been completed at least four (4) weeks before enrollment in this study (6 weeks for mitomycin-C or nitrosourea)
* Patients have recovered from the acute side effects due to prior therapy
* Life expectancy of > 3 months
* World Health Organization (WHO) Performance Status 0-2
* 18 years of age or older
* Adequate organ function as defined in the protocol

Exclusion Criteria:

* Prior therapy with CAMPATH
* Use of an investigational agent within two (2) weeks prior to study enrollment
* History of anaphylaxis following exposure to humanized monoclonal antibodies
* Known human immunodeficiency virus (HIV) positive
* Prior autologous bone marrow or stem cell transplant if within six (6) months of study entry
* A history or prior allogenic bone marrow transplant or organ transplant
* Known, symptomatic central nervous system (CNS) involvement with lymphoma
* Pregnant or lactating women
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (excluding skin infection, lower urinary tract infection, or oral infection), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2003-12; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (2):
- United States (2):
  - Duluth, Minnesota
  - Durham, North Carolina